CLINICAL TRIAL: NCT01765361
Title: Assessment of Ocrelizumab (OCR) Treatment Effects on Functional Impairment of MS Patients Enrolled in the Phase III Orchestra Programme Using Multimodal Evoked Potentials (EP) and Highresolution Electroencephalography (EEG)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EP-OCR
Record Dates: First submitted 2012-12-21; First posted 2013-01-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple Sclerosis (MS) is not only an 'inflammatory' demyelinating disease, but also includes axonal and neuronal injury in the grey matter . Neurodegenerative processes are partly independent of lesion formation and relapse activity , but represent the direct driver of clinical long-term disability and cognitive decline.

Multimodal evoked potentials (EP), i.e. the combination of visual, somato-sensory and motor EP (VEP, SSEP, MEP) have been shown prospectively to provide objective, monovectorial, and numerical data which are closely correlated to the EDSS. As EP capture the functional integrity of the examined systems they represent a method unbiased for directional changes, while remaining specific for the neuronal function, and hence can measure deterioration, as well as improvement, a germane advantage to capture drug response.

High-resolution electroencephalography (EEG) allow for explorative analysis of potential surrogate markers for cognitive decline.

Ocrelizumab (OCR), a humanized anti-CD20 monoclonal antibody has shown strong treatment effects on number of T1Gd-enhancing lesions , on new T1Gd-enhancing and new T2-hyperintense lesions as well as on the annualized relapse rate in a recent phase II trial in relapsing-remitting MS.

The present study will investigate the effects of OCR on multimodal evoked potentials (EP), Furthermore, quantitative EEG as a potential correlate of cognitive dysfunction and fatigue will be explored.

ELIGIBILITY:
Inclusion Criteria:

* definitive inclusion in one of the phase III trials on OCR: relapsing remitting multiple sclerosis (RRMS) patients in "Opera I" (WA21092B) or "Opera II" (WA21093), primary progressive multiple sclerosis (PPMS) patients in "Oratorio" (WA25046B) and fulfilling the respective inclusion criteria
* stable clinical state (at least 4 weeks after treatment with corticoids, when there was a relapse)
* Provision of written informed consent and ability to be compliant with the schedule of assessments of the present study

Exclusion Criteria:

* exclusion criteria of both phase III trials on OCR also apply to the present study
* additionally patients with movable metal implants, e.g. pace-maker, stents, deep brain stimulators are excluded; (patients with jaw- or bone-fixed metal implants can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a sub-sample of the above mentioned multi-center, randomized, double-blind, phase III trials ("Oratorio", "Opera I" and "Opera II") and will comprise approximately 100 PPMS and 100 RRMS patients. Treatment groups will only be disclosed after completion of the phase III trials.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
dΣ-EP | Baseline, 48 weeks, 96 weeks (RMS)/ Baseline, 48 weeks, 120 weeks (PPMS)
  The primary outcome measure is the change in the sum score of multimodal EP (dΣ-EP) after two years, which will be compared between treatment groups.

SECONDARY OUTCOMES:
d#-EP | Baseline, 48 weeks, 96 weeks (RMS)/ Baseline, 48 weeks, 120 weeks (PPMS)
  Secondary outcome measures are the change in number of abnormal EP (d#-EP) as well as change in cognitive performance and fatigue at two years.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, MD, Prof., Study Director — University Hospital, Basel, Switzerland
Locations (1):
- Dep. Neurology, Hospital of the University of Basel, Basel, Switzerland